CLINICAL TRIAL: NCT05830474
Title: Effect of Continuous Intra-airway Monitoring Under Visible Double-lumen Bronchial Catheter on Postoperative Complications of Lung Surgery (a Prospective, Single-center, Randomized, Controlled Clinical Study)
Brief Title: Effect of Continuous Intra-airway Monitoring Under Visible Double-lumen Bronchial Catheter on Postoperative Complications of Lung Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022YF060-01
Record Dates: First submitted 2023-01-31; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pulmonary Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (group T) (Experimental): lung isolation was performed with visual double-lumen bronchial catheter, andcontinuous airway monitoring and intervention were performed
  Interventions: Procedure: Continuous intra-airway monitoring and intervention during surgey
- Control group (group C) (No Intervention): lung isolation was performed with visual double-lumen bronchial catheter, and only intra-airway video was performed without monitoring

INTERVENTIONS:
Procedure: Continuous intra-airway monitoring and intervention during surgey — Continuous monitoring was performed by visual double lumen bronchial catheter. Once sputum or blood gushing into the tracheal carina was found in the distal bronchus on the surgical side, the above secretions were sucked out with a sputum suction tube under video monitoring until the removal was complete
  Arms: Test group (group T)

SUMMARY:
The incidence of postoperative pulmonary complications (PPCs) after thoracic surgery is as high as 30-50% [1-6], which is the main cause of postoperative morbidity, death and prolonged hospital stay. Optimization of risk factors in PPCs procedures is the focus of current research. Double lumen bronchial tube (DLT) is a commonly used lung isolation method for adult patients. It has the advantages of good lung isolation effect, sufficient exposure of the surgical field and easy to attract secretions in the airway. However, there are still some deficiencies in clinical precise positioning, long-term continuous detection during operation, early detection of catheter displacement and other emergencies. Continuous intra-airway monitoring is the main advantage of visual double-lumen bronchial catheter. It can quickly and easily determine the position of the catheter and quickly adjust the displacement, and timely and effectively clean up the secretion in the airway, which is conducive to the analysis and treatment of intraoperative hypoxemia. Whether these potential advantages can reduce the incidence of PPCs deserves our in-depth discussion. The research group randomly divided the patients who were scheduled to undergo thoracoscopic radical resection of lung cancer in the Union Hospital affiliated to Fujian Medical University into the test group (lung isolation with visible double-lumen bronchial catheter, continuous intra-airway monitoring and intervention) and the control group: (Pulmonary isolation was performed with visual double-lumen bronchial catheter, and only intra-airway video was performed without monitoring. The effect of continuous intra-airway monitoring under visual double-lumen bronchial catheter on postoperative complications of lung surgery was evaluated by Melbourne evaluation scale.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-80 years, BMI 18.5-28 kg/m2, male or female
* 2. Patients who are to undergo unilateral thoracoscopic resection of more than three lung segments or lobectomies
* 3. Patients who can be extubated with 35# and 37# double-lumen bronchial catheters after pre-anesthetic evaluation
* 4. Subjects voluntarily sign the informed consent form for this trial.
* 5. Patients or their caregivers are able to fill out the survey form and can correctly understand and cooperate with the postoperative rehabilitation instructions of the medical staff.
* 6. Patients have SPO2 ≥ 96% when inhaling air preoperatively

Exclusion Criteria:

* 1. Patients with limited ability to cooperate with the study, such as the presence of cognitive dysfunction, mental illness, speech impairment or severe visual impairment or hearing impairment
* 2.ASA ≥IV
* 3. difficult airway, abnormal tracheal development, main airway stenosis, tumor, tracheoesophageal fistula
* 4. Complex sleeve pneumonectomy, unilateral total pneumonectomy, bilateral lung surgery
* 5. Preoperative anemia, Hb≤100g/L
* 6. Serum albumin ≤ 35g/L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of pulmonary complications | 3 days after operation
  Evaluation of the incidence of pulmonary complications three days after surgery by the Melbourne Assessment Scale Melbourne Group Scale（Minimum value 0 points ；Max 8 points
  1. Oral temperature > 38°C;
  2. White blood cell count > 11.2×10^12/L or use respiratory antibiotics (except prophylactic antibiotics);
  3. Pneumonia or pulmonary infection diagnosed by the treating doctor;
  4. Chest X-ray examination suggested atelectasis or consolidation;
  5. Purulent sputum (yellow/green) with characteristics different from those before operation;
  6. Sputum microbiological examination was positive;
  7. Oxygen saturation of finger pulse < 90% under suction condition;
  8. Readmission or ICU stay > 36h due to respiratory problems
  If 4 or more of the above 8 items are satisfied, the subject is considered to have developed pulmonary complications.

SECONDARY OUTCOMES:
Double lumen tube displacement | during the operation
  The number of times that fiberoptic bronchoscopy should be used to check or adjust the position during the operation, the rate of displacement, the degree of displacement, the number and time of operation suspension due to the adjustment of the position of double-lumen tube, etc Position adjustment assisted by fiberoptic（Check only unadjusted available at the back □ mark ×）
  □NO : 1stTime：|__|__|min|__|__|second；□ 2stTime：|__|__|min|__|__|second：□ 3stTime：|__|__|min|__|__|second：□
  □YES： 1stTime：|__|__|min|__|__|second；□ 2stTime：|__|__|min|__|__|second：□ 3stTime：|__|__|min|__|__|second：□
Intubation effectiveness | during the operation
  Time taken for successful intubation and positioning (time from laryngoscope exposure to successful positioning of double lumen bronchial tube), success rate of first intubation and positioning, and probability of using fiber bronchoscopy for positioning
  1. Number of intubation times:|__| Times
  2. Time taken for successful intubation positioning:|__|__| Minutes|__|__| seconds
  3. Whether fiber bronchoscopy is used for positioning: □ No □ Yes
Hypoxemia during operation | during the operation
  Intraoperative SPO2<90%
  □ Yes □ No
  1. st time:|__|__| Minutes|__|___| Seconds;
  2. nd time:|__|__| Minutes|__|___| Seconds;
  3. rd time:|__|__| Minutes|__|___| Seconds;
Intraoperative carbon dioxide accumulation | during the operation
  PaCO2>45mmHg：□ No □ Yes: Duration|__|__| Minutes|__|__| Seconds;
Incidence of tracheal intubation complications | three days after operation
  Incidence of postoperative sore throat, hoarseness, etc.
Lung atrophy quality | during the operation
  Lung atrophy quality during the operation（The condition is judged by the thoracic surgeon）
  口Excellent visual field exposure, complete collapse of lung 口Medium The lungs are basically collapsed, but there's still residual air 口Poor Partial collapse or even non-collapse of the lung requires surgical intervention to expose the visual field
Effectiveness of sputum suction | Postoperative
  1. Postoperative video review: The suction rate during intraoperative sputum suction:
     □ 80%-100%； □ 50-80%; □ 0-50%;
  2. After tracheal extubation, take photos to compare the secretion at the end of the bronchus:
     * None
     * Yes: □ Small amount (secretions adhering to the wall less than 2cm); □ Moderate amount (secretion adhering to the wall 2-4cm); □ Large amount (secretions sticking to the wall exceeding 4cm)

IPD SHARING:
Plan to Share IPD: Undecided